CLINICAL TRIAL: NCT06889142
Title: Proof-of-Concept Study: Investigating the Impact of NMN Supplementation on CD4+ T Cell Recovery in Virologically Suppressed HIV Patients With Immunological Failure
Brief Title: Impact of NMN Supplementation on CD4+ T Cell Recovery in HIV Patients With Immunological Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Collaborators: DoNotAge.org (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-089
Record Dates: First submitted 2025-03-03; First posted 2025-03-21 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; immunologic failure; proof of concept; CD4+ T cell recovery; immunological non-responders; Nicotinamide Mononucleotide
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Nicotinamide Mononucleotide

STUDY DESIGN:
Intervention Model Description: proof of concept
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with 1,000mg Nicotinamide Mononucleotide daily (Experimental)
  Interventions: Dietary Supplement: Nicotinamide Mononucleotide

INTERVENTIONS:
Dietary Supplement: Nicotinamide Mononucleotide — The dietary supplement NMN [1,000mg] will be taken orally by participants daily for a total of 12 weeks
  Other Names: NMN

SUMMARY:
This proof-of-concept study aims to investigate the potential impact of supplementing with Nicotinamide Mononucleotide (NMN), a direct precursor of NAD+ on CD4+ T cell recovery in virologically suppressed HIV patients experiencing immunological failure on ART. We hypothesize that NMN supplementation will increase intracellular NAD+ levels, thereby improving CD4+ T cell function and potentially reversing immunological failure. A small cohort of patients will be recruited to evaluate the primary outcome of change in CD4+ T cell count from baseline to the end of the study period after receiving NMN daily for 12 weeks. Secondary outcomes including safety and tolerability, impact on pro-inflammatory markers, increase in NAD+ levels, immune activation markers and change in quality of life questionnaire scores. Patients will participate in two in person visits including a baseline and end of study with two telephone encounters. Patients will take 1,000mg NMN daily for a total of 12 weeks during which they will keep a daily log of doses taken and any side effects experienced. At all visits labs and quality of life questionnaire will be completed with complete physical exam to be done at baseline and end of study visit.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected adults aged 18 years or older
* Virologically suppressed on ART documented with two negative viral loads separated by at least 6 months
* Confirmed diagnosis of immunological failure (CD4+ T cell count <350 cells/µL 2 years after effective ART initiation)
* Willing to provide informed consent

Exclusion Criteria:

* Active opportunistic infections
* Known allergies or sensitivities to NMN or any components of the NMN supplement
* Current or recent use of other supplements or medications known to affect NAD+ metabolism (Niacin, NR, NMNH, etc.)
* Pregnancy or breastfeeding
* Significant liver or kidney disease
* Active malignancy
* History of uncontrolled substance abuse
* Severe medical conditions that might interfere with study participation
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 12 weeks
  The primary outcome of this study will be the change in CD4+ T cell count from baseline to the end of the study period. [normal range: 500-1500 cells/mm^3; improved outcomes with increase to normal range]

SECONDARY OUTCOMES:
CD38 | collected at baseline visit followed by monthly collections for total of 3 months
  Changes in immune activation markers - CD38 expression [healthy individuals expression on T cell <10-20%, untreated HIV elevated >60-90%, HIV on ART ~ 20-30%; low percentage correlates with improved immune function]
HLA-DR expression | collected at baseline visit followed by monthly collections for total of 3 months
  HLA-DR expression [healthy individuals <5-10% HLA DR CD 4+ T cell expression and <5%
TNF-alpha | collected at baseline visit followed by monthly collections for total of 3 months
  (Ref Interval: <=7.2) Cytokines- Results are used to understand the pathophysiology of immune, infectious, or inflammatory disorders
NAD(+) levels | collected at baseline visit followed by monthly collections for total of 3 months
  Ranges from 10-500 µM during normal physiological state; however, it's levels can vary by age as well as metabolic and disease states
IL-6 | collected at baseline visit followed by monthly collections for total of 3 months
  (Ref Interval: <=2.0 pg/mL ) Cytokines- Results are used to understand the pathophysiology of immune, infectious, or inflammatory disorders
HS-CRP | collected at baseline visit followed by monthly collections for total of 3 months
  Ref Interval: <=3.0 mg/L
Changes on Quality-of-life Questionnaire (QOL): WHO QOL HIV BREF | collected at baseline visit followed by monthly collections for total of 3 months
  Domain scores between 4-20 with higher score correlating with improved QOL

CONTACTS AND LOCATIONS:
Overall Officials: Madelyn Mirande, DO, Study Chair — TriHealth Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shi H, Enriquez A, Rapadas M, Martin EMMA, Wang R, Moreau J, Lim CK, Szot JO, Ip E, Hughes JN, Sugimoto K, Humphreys DT, McInerney-Leo AM, Leo PJ, Maghzal GJ, Halliday J, Smith J, Colley A, Mark PR, Collins F, Sillence DO, Winlaw DS, Ho JWK, Guillemin GJ, Brown MA, Kikuchi K, Thomas PQ, Stocker R, Giannoulatou E, Chapman G, Duncan EL, Sparrow DB, Dunwoodie SL. NAD Deficiency, Congenital Malformations, and Niacin Supplementation. N Engl J Med. 2017 Aug 10;377(6):544-552. doi: 10.1056/NEJMoa1616361. PMID 28792876
- [Background] Braidy N, Berg J, Clement J, Khorshidi F, Poljak A, Jayasena T, Grant R, Sachdev P. Role of Nicotinamide Adenine Dinucleotide and Related Precursors as Therapeutic Targets for Age-Related Degenerative Diseases: Rationale, Biochemistry, Pharmacokinetics, and Outcomes. Antioxid Redox Signal. 2019 Jan 10;30(2):251-294. doi: 10.1089/ars.2017.7269. Epub 2018 May 11. PMID 29634344
- [Background] Song Q, Zhou X, Xu K, Liu S, Zhu X, Yang J. The Safety and Antiaging Effects of Nicotinamide Mononucleotide in Human Clinical Trials: an Update. Adv Nutr. 2023 Nov;14(6):1416-1435. doi: 10.1016/j.advnut.2023.08.008. Epub 2023 Aug 22. PMID 37619764
- [Background] Lebouche B, Jenabian MA, Singer J, Graziani GM, Engler K, Trottier B, Thomas R, Brouillette MJ, Routy JP. The role of extended-release niacin on immune activation and neurocognition in HIV-infected patients treated with antiretroviral therapy - CTN PT006: study protocol for a randomized controlled trial. Trials. 2014 Oct 7;15:390. doi: 10.1186/1745-6215-15-390. PMID 25293882
- [Background] Mo Y, Yue M, Yim LY, Zhou R, Yu C, Peng Q, Zhou Y, Luk TY, Lui GC, Huang H, Lim CYH, Wang H, Liu L, Sun H, Wang J, Song Y, Chen Z. Nicotinamide mononucleotide impacts HIV-1 infection by modulating immune activation in T lymphocytes and humanized mice. EBioMedicine. 2023 Dec;98:104877. doi: 10.1016/j.ebiom.2023.104877. Epub 2023 Nov 17. PMID 37980794
- [Background] MD MG. Unveiling the Nexus of CD38 Overactivation, NAD+ Depletion, and Mitochondrial Dysfunction in Immunological Failure Among Virologically Suppressed HIV Patients. 2024(https://nortonhealthcaremedicaljournal.scholasticahq.com/article/118564-unveiling-the-nexus-of-cd38-overactivation-nad-depletion-and-mitochondrial-dysfunction-in-immunological-failure-among-virologically-suppressed-hiv).
- [Background] Zhu A, Real F, Zhu J, Greffe S, de Truchis P, Rouveix E, Bomsel M, Capron C. HIV-Sheltering Platelets From Immunological Non-Responders Induce a Dysfunctional Glycolytic CD4+ T-Cell Profile. Front Immunol. 2022 Feb 11;12:781923. doi: 10.3389/fimmu.2021.781923. eCollection 2021. PMID 35222352
- [Background] Fan L, Li P, Yu A, Liu D, Wang Z, Wu Y, Zhang D, Zou M, Ma P. Prevalence of and prognosis for poor immunological recovery by virally suppressed and aged HIV-infected patients. Front Med (Lausanne). 2023 Oct 19;10:1259871. doi: 10.3389/fmed.2023.1259871. eCollection 2023. PMID 37928477
- [Background] Dessie G, Mulugeta H, Wagnew F, Zegeye A, Kiross D, Negesse A, Aynalem YA, Getaneh T, Ohringer A, Burrowes S. Immunological Treatment Failure Among Adult Patients Receiving Highly Active Antiretroviral Therapy in East Africa: A Systematic Review and Meta-Analysis. Curr Ther Res Clin Exp. 2021 Jan 5;94:100621. doi: 10.1016/j.curtheres.2020.100621. eCollection 2021. PMID 34306262
- [Background] Carvalho-Silva WHV, Andrade-Santos JL, Souto FO, Coelho AVC, Crovella S, Guimaraes RL. Immunological recovery failure in cART-treated HIV-positive patients is associated with reduced thymic output and RTE CD4+ T cell death by pyroptosis. J Leukoc Biol. 2020 Jan;107(1):85-94. doi: 10.1002/JLB.4A0919-235R. Epub 2019 Nov 5. PMID 31691351
- [Background] Burnie J, Fernandes C, Chaphekar D, Wei D, Ahmed S, Persaud AT, Khader N, Cicala C, Arthos J, Tang VA, Guzzo C. Identification of CD38, CD97, and CD278 on the HIV surface using a novel flow virometry screening assay. Sci Rep. 2023 Dec 27;13(1):23025. doi: 10.1038/s41598-023-50365-0. PMID 38155248
- [Background] Bono V, Augello M, Tincati C, Marchetti G. Failure of CD4+ T-cell Recovery upon Virally-Effective cART: an Enduring Gap in the Understanding of HIV+ Immunological non-Responders. New Microbiol. 2022 Jul;45(3):155-172. PMID 35920870